CLINICAL TRIAL: NCT01280058
Title: A 2-arm Randomized Phase II Study of Carboplatin, Paclitaxel Plus Reovirus Serotype-3 Dearing Strain (Reolysin) vs. Carboplatin and Paclitaxel in the First Line Treatment of Patients With Recurrent or Metastatic Pancreatic Cancer
Brief Title: Carboplatin and Paclitaxel With or Without Viral Therapy in Treating Patients With Recurrent or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02567; NCI-2011-02567 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OSU 10045; OSU-10045; CDR0000692060; 8601 (Other: Ohio State University Comprehensive Cancer Center); 8601 (Other: CTEP); N01CM00070 (NIH); N01CM62207 (NIH); P30CA016058 (NIH)
Record Dates: First submitted 2011-01-18; First posted 2011-01-20 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Pancreatic Acinar Cell Carcinoma; Pancreatic Ductal Adenocarcinoma; Recurrent Pancreatic Carcinoma; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Carboplatin; Paclitaxel; Taxes; reolysin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (wild-type reovirus, carboplatin, paclitaxel) (Experimental): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1 and wild-type reovirus IV over 60 minutes on days 1-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Biological: Wild-type Reovirus
- Arm II (carboplatin, paclitaxel) (Experimental): Patients receive paclitaxel and carboplatin as in Arm I. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may crossover to Arm I.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplat; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Biological: Wild-type Reovirus — Given IV
  Other Names: Reolysin
  Arms: Arm I (wild-type reovirus, carboplatin, paclitaxel)

SUMMARY:
This phase II trial studies how well carboplatin and paclitaxel with or without viral therapy works in treating patients with pancreatic cancer that has come back or has spread to other places in the body. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Viral therapy may be able to kill tumor cells without damaging normal cells. It is not yet known whether carboplatin and paclitaxel are more effective with or without viral therapy in treating pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the improvement in progression-free survival with Reolysin (wild-type reovirus), carboplatin, and paclitaxel relative to carboplatin and paclitaxel alone in patients with recurrent or metastatic pancreatic cancer.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of Reolysin in combination with carboplatin and paclitaxel versus without Reolysin in patients with recurrent or metastatic pancreas cancer.

II. To compare the treatment groups for other efficacy endpoints such as overall response rate and overall survival.

III. To define how the combination of Reolysin and carboplatin and paclitaxel (CP) modulate factors regulating immunity to reovirus and its persistence in the system circulation of patients with pancreatic cancer.

IV. To prospectively establish and validate the relationship between Ras mutations in tumor samples and response to Reolysin.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive paclitaxel intravenously (IV) over 3 hours and carboplatin IV over 30 minutes on day 1 and wild-type reovirus IV over 60 minutes on days 1-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive paclitaxel and carboplatin as in Arm I. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may crossover to Arm I.

After completion of study treatment, patients are followed up at 1 month and then every 2 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the pancreas that is recurrent or metastatic; cytological confirmation is not allowed on this study; paraffin embedded tissue from tumor blocks will be required from patients before enrolling on this study; diagnosis of pancreas cancer with histologic confirmation of adenocarcinoma would suffice
* Patients must have measurable disease, defined as one lesion that can be accurately measured in at least one dimension per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 (longest diameter to be recorded) as >= 10 mm by spiral computed tomography (CT) scan (CT scan slice thickness no greater than 5 mm); malignant lymph nodes will be considered measurable if they are >= 15 mm in short axis; for patients previously irradiated, the measurable lesion must be outside the radiated field
* Patients must not have received any prior chemotherapy in metastatic setting; patients who have received prior chemotherapy in the adjuvant setting will not be eligible for our study; patients should not have received prior Reolysin; prior palliative radiation therapy or major surgery must have occurred at least 28 days prior to study enrollment; prior minor surgeries (such as laparoscopies) must have occurred at least 14 days prior to study enrollment; prior minor procedures such as biopsies and mediport placement must have occurred at least 48 hours prior to study enrollment
* Eastern Cooperative Oncology Group (ECOG) status =< 1 (Karnofsky >= 70%)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L International System of Units (SI) units
* Platelet count >= 100 x10^9/L SI units
* Hemoglobin >= 8.5 g/dL SI units
* Serum creatinine =< 1.5 mg/dL OR creatinine clearance >= 60 mL/min
* Bilirubin =< upper limit of normal (ULN) (=< 2 x ULN if it is non-rising for a period of 10 days prior to initiation of therapy)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 X ULN
* Troponin I < ULN
* All patients must have signed an informed consent indicating that they are aware of the neoplastic nature of their disease and have been informed of the procedures of the protocol, the experimental nature of the therapy, alternatives, potential benefits, side effects, risks, and discomforts
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; patients must be able to avoid direct contact with pregnant or nursing women, infants and immunocompromised individuals while on study and for >= 3 weeks following the last dose of Reolysin administration
* All patients must be willing and able to comply with scheduled visits, the treatment plan, and laboratory tests

Exclusion Criteria:

* Patients may not be receiving any other investigational agents or concurrent therapy with other anti-cancer agents while on study
* Patients with untreated brain metastases will be excluded from this clinical trial; however, patients with resected oligometastasis are eligible if postresection magnetic resonance imaging (MRI) demonstrates resolution; gamma-knife treated patients are also eligible if there are no more than two treated metastases confined to the same area of the brain and a post treatment MRI shows a decrease in the metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Reolysin or other agents used in the study
* Patients may not have received any viral-based therapy within the past 6 months
* Patients must have NO continuing acute toxic effects (except alopecia) of any prior radiotherapy, chemotherapy, or surgical procedures; all such effects must have resolved to Common Terminology Criteria for Adverse Events (CTCAE, version [v.] 4 ) grade =< 1 prior to study enrollment
* Patients must not have grade 2 or higher baseline peripheral neuropathy according to CTCAE v. 4
* Patients with uncontrolled cardiac dysfunction or arrhythmia, including a myocardial infarction in the preceding 6 months, known cardiac ejection fraction < 40%, symptomatic congestive heart failure, or unstable angina pectoris
* Patients must not be receiving concurrent systemic immunosuppressive therapy
* Patients must not have known human immunodeficiency virus (HIV) infection or active hepatitis B or C
* Patients must not have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or known psychiatric illness/social situations that would limit compliance with study requirements
* Patients must not have dementia or altered mental status that would prohibit informed consent
* Patients must not have other known severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation, study drug administration, or may interfere with the interpretation of study results that, in the judgment of the Principal Investigator, would make the patient inappropriate for this study
* Pregnant women are excluded from this study; breastfeeding should be discontinued while the mother is being treated with the agents in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2016-01-19 (Actual); Study Completion 2016-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Noonan, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (6):
- United States (6):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma

REFERENCES:
- [Result] Noonan AM, Farren MR, Geyer SM, Huang Y, Tahiri S, Ahn D, Mikhail S, Ciombor KK, Pant S, Aparo S, Sexton J, Marshall JL, Mace TA, Wu CS, El-Rayes B, Timmers CD, Zwiebel J, Lesinski GB, Villalona-Calero MA, Bekaii-Saab TS. Randomized Phase 2 Trial of the Oncolytic Virus Pelareorep (Reolysin) in Upfront Treatment of Metastatic Pancreatic Adenocarcinoma. Mol Ther. 2016 Jun;24(6):1150-1158. doi: 10.1038/mt.2016.66. Epub 2016 Apr 4. PMID 27039845
- [Derived] Farren MR, Mace TA, Geyer S, Mikhail S, Wu C, Ciombor K, Tahiri S, Ahn D, Noonan AM, Villalona-Calero M, Bekaii-Saab T, Lesinski GB. Systemic Immune Activity Predicts Overall Survival in Treatment-Naive Patients with Metastatic Pancreatic Cancer. Clin Cancer Res. 2016 May 15;22(10):2565-74. doi: 10.1158/1078-0432.CCR-15-1732. Epub 2015 Dec 30. PMID 26719427

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized between February 2011 and April 2014
Groups:
- Arm A (Wild-type Reovirus, Carboplatin, Paclitaxel): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1 and wild-type reovirus IV over 60 minutes on days 1-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Carboplatin: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Paclitaxel: Given IV
  Wild-type Reovirus: Given IV
- Arm B (Carboplatin, Paclitaxel): Patients receive paclitaxel and carboplatin as in Arm I. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may crossover to Arm I.
  Carboplatin: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Paclitaxel: Given IV
Period: Overall Study
Arm/Group | Arm A (Wild-type Reovirus, Carboplatin, Paclitaxel) | Arm B (Carboplatin, Paclitaxel)
Started | 36 | 37
Completed | 36 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Wild-type Reovirus, Carboplatin, Paclitaxel) | Arm B (Carboplatin, Paclitaxel) | Total
Number analyzed (Participants) | 36 | 37 | 73
Age, Continuous [Median (Full Range); unit: years] | 61.5 [39 to 84] | 66 [45 to 81] | 64 [39 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 32
  Male | 22 | 19 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 32 | 35 | 67
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 37 | 73

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Using RECIST v. 1.1
Description: The progression-free survival distributions between the two arms will be compared using log-rank tests. Progression-free survival curves will be constructed using the Kaplan-Meier product limit method, and additional analyses will be done using the Cox proportional hazards model.
Time Frame: From study entry to the date of documented progression and/or death, assessed up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Wild-type Reovirus, Carboplatin, Paclitaxel) | Arm B (Carboplatin, Paclitaxel)
Number analyzed (Participants) | 36 | 37
months | 4.9 [3.0 to 6.3] | 5.2 [2.3 to 6.2]

2. Secondary Outcome: Incidence of Severe (Grade 3+) Adverse Events That Are Classified as Either Possibly, Probably, or Definitely Related to Study Treatment, as Assessed by NCI CTCAE Version 4.0
Description: Toxicities will be described for each treatment arm, but will also be compared between the arms. Fisher's exact tests will be used to quantitatively compare the incidence of severe as well as specific toxicities of interest between the treatment arms and we will graphically assess differences in maximum grades observed for toxicities between the arms.
Time Frame: Up to 4 years
Measure: Number; unit: percentage of patients
Arm/Group | Arm A (Wild-type Reovirus, Carboplatin, Paclitaxel) | Arm B (Carboplatin, Paclitaxel)
Number analyzed (Participants) | 36 | 37
percentage of patients
  Neutropenia | 56 | 59
  Leukopenia | 33 | 46
  Thrombocytopenia | 28 | 24
  Anemia | 25 | 30
  Febrile Neutropenia | 8 | 11
  Fatigue | 11 | 8
  Infection | 11 | 5
  Dose Delay | 37 | 54
  Dose reduction | 36 | 43

3. Secondary Outcome: Overall Response Rate (Partial or Complete Response) Evaluated Using the Standard RECIST v. 1.1
Description: 95% confidence intervals will be calculated. Differences in objective response rates between the treatment arms will be assessed using Fisher's exact test.
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Wild-type Reovirus, Carboplatin, Paclitaxel) | Arm B (Carboplatin, Paclitaxel)
Number analyzed (Participants) | 36 | 37
Participants
  Partial Response | 7 | 7
  Complete Response | 0 | 0

4. Secondary Outcome: Overall Survival
Description: Evaluated and compared between the two treatment groups using log-rank statistics and graphically using the methods of Kaplan and Meier.
Time Frame: From study entry to the time of death due to any cause, assessed up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Wild-type Reovirus, Carboplatin, Paclitaxel) | Arm B (Carboplatin, Paclitaxel)
Number analyzed (Participants) | 36 | 37
months | 7.3 [4.8 to 11.2] | 8.8 [6.6 to 11.8]

5. Other Pre Specified Outcome: Immunologic Correlative Markers
Description: The inflammatory cytokine profile, immune effector cell phenotype and function, and NARA titers will be assessed and compared. Patterns of change in the longitudinal data on these markers will be evaluated for each of the correlative outcomes of interest.
Time Frame: Up to day 1 of course 12
Population: data was not collected
Arm/Group | Arm I (Wild-type Reovirus, Carboplatin, Paclitaxel) | Arm II (Carboplatin, Paclitaxel)
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Percentage of Patients With Ras Pathway Activation
Description: The 95% confidence interval will be assessed. Cochran-Mantel-Haenszel test will be used to assess differences in the relationships between response and Ras pathway activation and the association of treatment groups on these relationships.
Time Frame: Baseline
Measure: Number; unit: percentage of patients
Arm/Group | Arm A (Wild-type Reovirus, Carboplatin, Paclitaxel) | Arm B (Carboplatin, Paclitaxel)
Number analyzed (Participants) | 36 | 37
percentage of patients | 71 | 75

ADVERSE EVENTS:
Description: The National Cancer Institutes (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 was used for adverse event grading and reporting.
Groups:
- Arm A (Wild-type Reovirus, Carboplatin, Paclitaxel): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1 and wild-type reovirus IV over 60 minutes on days 1-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Carboplatin and Paclitaxel were given IV. Wild-type Reovirus: Given IV
- Arm B (Carboplatin, Paclitaxel): Patients receive paclitaxel and carboplatin as in Arm I. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may crossover to Arm I. Carboplatin and Paclitaxel were given IV
Arm/Group | Arm A (Wild-type Reovirus, Carboplatin, Paclitaxel) | Arm B (Carboplatin, Paclitaxel)
Serious Adverse Events (participants affected / at risk) | 36/36 | 37/37
Other Adverse Events (participants affected / at risk) | 36/36 | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Wild-type Reovirus, Carboplatin, Paclitaxel) (N=36) | Arm B (Carboplatin, Paclitaxel) (N=37)
Anemia (Blood and lymphatic system disorders) | 10 (10) | 11 (11)
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain-cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 5 (5)
Ascites (Gastrointestinal disorders) | 3 (3) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestional hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (7) | 7 (7)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 4 (4)
Edema limbs (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 6 (6) | 2 (2)
Fever (General disorders) | 1 (1) | 1 (1)
Infusion related reaction (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 2 (2) | 3 (3)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Infections (Infections and infestations) | 2 (2) | 2 (2)
Lung Infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Skin Infection (Infections and infestations) | 2 (2) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 2 (2)
Blood bilirubin increased (Investigations) | 7 (7) | 4 (4)
Cardiac troponin I increaesd (Investigations) | 3 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 15 (15) | 13 (13)
Platelet count decreased (Investigations) | 10 (10) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
White blood cell decreased (Investigations) | 10 (10) | 8 (8)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Peripheral sensory (Nervous system disorders) | 2 (2) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 2 (2) | 0 (0)
Confusion (Psychiatric disorders) | 4 (4) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypostension (Vascular disorders) | 1 (1) | 2 (2)
Thromboembolic event (Vascular disorders) | 4 (4) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Wild-type Reovirus, Carboplatin, Paclitaxel) (N=36) | Arm B (Carboplatin, Paclitaxel) (N=37)
Neutropenia (Blood and lymphatic system disorders) | 20 (20) | 22 (22)
Leukopenia (Blood and lymphatic system disorders) | 12 (12) | 17 (17)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (10) | 9 (9)
Anemia (Blood and lymphatic system disorders) | 9 (9) | 11 (11)
Febrile Neutropenia (Infections and infestations) | 3 (3) | 4 (4)
Fatigue (General disorders) | 4 (4) | 3 (3)
Infection (Infections and infestations) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less